CLINICAL TRIAL: NCT04653818
Title: Does Directly Acting Antivirals Usage Affect HCV Related Hepatocellular Carcinoma Recurrence After Percutaneous Ablation: A Randomized Controlled Trial
Brief Title: HCV Related Hepatocellular Carcinoma Recurrence After Directly Acting Antivirals: A Randomized Controlled Trial
Acronym: RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Kamal, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0304763
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma; Hepatitis C; Neoplasm Recurrence; Treatment Complication
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C; Recurrence | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: masking for radiologists who assess HCC recurrence only. Patients and physicians: not masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAAs group (Active Comparator): Those with complete HCC ablation who will start sofosbuvir / velpatasvir aiming to eradicate HCV.
  Interventions: Drug: Velpatasvir/Sofosbuvir
- Postponed DAAs group (Active Comparator): Those who will not start DAAs within the 12 months follow up from HCC ablation procedure. Patients of this group will receive DAAs provided that there is no HCC recurrence after the end of 1 year.
  Interventions: Drug: Velpatasvir/Sofosbuvir

INTERVENTIONS:
Drug: Velpatasvir/Sofosbuvir — sofosbuvir / velpatasvir will be given for 12 weeks aiming to eradicate HCV. Ribavirin will be added for Child-Pugh B patients or treatment will be extended for 24 weeks for those who are Ribavirin intolerant.

SUMMARY:
Data regarding hepatocellular carcinoma (HCC) recurrence after directly acting antivirals (DAAs) given for hepatitis C virus treatment are contradictory. Surprisingly, some studies reported that DAAs are accompanied with higher HCC recurrence. But, other studies showed no rise or even decrease in HCC recurrence. Most of these studies were retrospective and some were non-randomized prospective studies. Here investigators aim to perform a randomized controlled trial to study this issue.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh A and B subjects with hepatitis C related < 5 cm single or up to 3 hepatocellular carcinomas without any vascular or extrahepatic involvement

Exclusion Criteria:

* Those with positive HBsAg, history of alcohol consumption, patients with other known causes of chronic liver disease, patients who have received previous DAAs for HCV and patients who have received previous locoregional treatment for HCC will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
HCC recurrence | 1 year after HCC ablation procedure

SECONDARY OUTCOMES:
changes in Child-Pugh scores over time | 1 year from HCC ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kamal, MD, PhD, Principal Investigator — Lecturer of Internal Medicine and Hepatology, Faculty of Medicine, Alexandria University
Locations (1):
- Alexandria University, Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kamal A, Metawea M, Omar H, Ghallab M, Kassem A, Naguib H. Hepatitis C Virus-Related One-Year Hepatocellular Carcinoma Recurrence After Directly Acting Antivirals: A Randomized Controlled Trial. J Gastrointest Cancer. 2024 Jun;55(2):913-923. doi: 10.1007/s12029-024-01035-5. Epub 2024 Mar 4. PMID 38436921